

## Evaluation of Seismocardiography (SCG) as a viable tool in assessing fitness in Oesophago-Gastric surgery



IRAS ID: 343434 Centre number: TBC Study number: TBC

Participant Identification Number for this trial: TBC

## **CONSENT FORM**

Title of project: Evaluation of Seismofit® as a viable tool in assessing fitness in Oesophago-Gastric surgery Name of researcher: Mr Andrew Davies

| | | Please<br>initial<br>box |
|---|---|---|
| 1. | I confirm that I have read the information sheet dated (version) for the above study. I have had the opportunity to think about the information, ask questions and have had helpful answers that I am happy with. | |
| 2. | I understand that my participation is voluntary and that I can withdraw at any time without giving a reason, and without my medical care or legal rights being affected. | |
| 3. | I give permission for the research team to access my medical records for the purposes of this research study. I understand that my anonymised data will be transferred to the Commercial company Ventriject and may be used to improve the Seismofit algorithm in the future. I understand that should an improved algorithm be generated from this study; this algorithm may be used in commercial purposes in the future. | |
| 4. | I understand that should an improved algorithm be generated from this study; this algorithm may be used in commercial purposes in the future. | |
| 5. | I understand that relevant sections of my medical notes and data collected during the study, may be looked at by individuals from the Sponsor (Guy's and St Thomas' NHS Foundation Trust and/or King's College London), from regulatory authorities or from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these people to have access to my data and medical records | |
| 6. | I give permission for my personal information (including <i>date of birth</i> ) to be passed to King's College London so that I can take part in of the study | |
| 7. | I understand that data collected about me during the study may have identifying details removed to convert it into pseudonymised or anonymised data. | |
| 8. | I agree to take part in the above study | |
| 9. | If at the end of the study, you would like to receive information on the results of the study, please provide an email address below. On completion of this study, we can send you a summary of the results of this study should you wish to have this. | |

When completed: 1 for participant; 1 for researcher site file; 1 to be kept in medical notes.



## Evaluation of Seismocardiography (SCG) as a viable tool in assessing fitness in Oesophago-Gastric surgery



| | 10. If you would like to have the option to allow the research team to securely store your contact details and agree to be contacted about other ethically approved research studies, please initial the box on the right. | | |
|---|---|---|---|
| Name of Pa | articipant | Date | Signature |
| Email addr | ess if you wish to see | the results completion of the stu | |
| | , | ' | |
| Name of Petaking cons | | Date | Signature |

When completed: 1 for participant; 1 for researcher site file; 1 to be kept in medical notes.

IRAS: 342434 Version 2.0 (27/05/2025) Page2